CLINICAL TRIAL: NCT01009957
Title: Everolimus on CKD (Chronic Kidney Disease) Progression in ADPKD Patients
Brief Title: Everolimus on CKD Progression in ADPKD Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: After primary completition date, experimental drug was no longer available
Sponsor: A. Manzoni Hospital (Other)
Responsible Party: Principal Investigator, Prof. Francesco Locatelli, Prof. Francesco Locatelli, A. Manzoni Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PolEver
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Polycystic Kidney Diseases
Keywords: ADPKD; CKD; Renal disease progression; Everolimus
MeSH Terms: conditions — Polycystic Kidney Diseases; Polycystic Kidney, Autosomal Dominant | interventions — Everolimus; MTOR Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Experimental): Everolimus + standard therapy for CKD
  Interventions: Drug: Everolimus
- Control (No Intervention): Standard therapy for CKD

INTERVENTIONS:
Drug: Everolimus — 0.75 mg x 2 / day
  Other Names: mTOR inhibitors
  Arms: Everolimus

SUMMARY:
The study will evaluate whether the administration of everolimus (1.5 mg/day) can slow down the progression of CKD in ADPKD patients.

DETAILED DESCRIPTION:
Considering the inhibitor activity of Everolimus on mTOR, our hypothesis is to evaluate its possible utility on the progression of CKD in ADPKD patients by reducing the rate of increase of renal cysts.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects over 18 years of both genders
2. Clinical diagnosis of autosomal dominant polycystic kidney disease (ADPKD)
3. GFR, according to MDRD formula, between 30 and 90 ml/min/1.73 mq
4. Previous follow up of two years, with a creatinine evaluation at least once a year
5. GFR reduction of at least 2.5 ml/min/year (according to MDRD formula)

Exclusion Criteria:

1. Pregnancy, lactating, males and females without adequate contraception
2. Leucopenia (< 3,000 leucocytes/mm3) or thrombocytopenia (< 100,000 platelets/mm3)
3. Dyslipidemia (cholesterol or triglycerides > 260 mg/dl with treatment)
4. Urinary tract infection
5. Patients who cannot undergoing NMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-06; Primary Completion 2014-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reduction of GFR (according to MDRD formula) during a two-year follow up | Two year-followup

SECONDARY OUTCOMES:
reduction of creatinine clearance and GFR (according to Cockcroft-Gault formula) during a two-year follow up | Two year-followup
changes in kidney size and renal and liver cysts dimensions evaluated by NMR at basal and at the end of the study | Two year-followup
safety profile of everolimus (leucopenia, thrombocytopenia, lipid profile and other adverse events | Two year-followup
evaluation of phosphatemia, phosphaturia and urinary cytokines on primary end point | Two year-followup

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Locatelli, MD, Study Chair — Nephrology and Dialysis Department - A. Manzoni Hospital
Locations (7):
- Italy (7):
  - A.O. Spedali Civili Di Brescia, Brescia
  - Alessandro Manzoni Hospital, Nephrology and Dialysis Department, Lecco
  - Modena Hospital, Modena
  - Dipartimento di Patologia Sistematica - Università Federico 2°, Napoli
  - Ospedale "Guglielmo da Saliceto" - Nephrology and Dialysis Department, Piacenza
  - C.M.I.D. - Presidi Ospedalieri ASL 4, Torino
  - Ospedale Civile San Bortolo Vicenza, Vicenza